## **Statistical Analysis Plan**

## A Multicenter Study of the NEUWAVE Flex Microwave Ablation System in the Ablation of Medically Inoperable Primary Soft Tissue Lesions of the Lung: An Initial Experience

**Protocol Number: NEU 2017 06** 

Protocol Version: Amendment 2 (Version 3.0), 25JUL2018

This document is a confidential communication. The recipient agrees that no unpublished information contained herein will be published or disclosed without prior written approval. This document may be disclosed to the appropriate ethics committees or to duly authorized representatives of the U.S. Food and Drug Administration or other responsible regulatory authorities, under the condition that they are requested to keep it confidential.

SAP Version: 1.0 SAP Revision Date: 29JAN2020

## **Revision History**

| Version Number | Version Date | Reasons for Revision |
|----------------|--------------|----------------------|
| 1.0 | 29JAN2020 | Original Document |

#### **Table of Contents**

| 1 | Study Overview | 4 |
|---|---|---|
| | 1.1 Study Objectives | 4 |
| | 1.2 Study Design | 5 |
| 2 | Treatment Assignment | 5 |
| 3 | Randomization and Blinding Procedures | 5 |
| 4 | Interval Windows | 5 |
| 5 | Levels of Significance | 6 |
| 6 | Analysis Sets | 6 |
| 7 | Sample Size Justification | 6 |
| 8 | Data Safety Monitoring Board | 6 |
| 9 | Analyses to be Conducted | 7 |
| | 9.1 General Conventions | 7 |
| | 9.2 Disposition of Study Subjects | 7 |
| | 9.3 Demographic, Baseline, and Subject Health Status Characteristics | 7 |
| | 9.4 Primary Endpoint Analyses | |
| | 9.5 Secondary Endpoint Analyses | 8 |
| | 9.6 Safety Analyses | 8 |
| | 9.7 Additional Endpoint Analyses | 8 |
| | 9.8 Plans for Interim Analysis | 9 |
| | 9.9 Handling of Missing Data | 9 |
| | 9.10 Sensitivity Analyses | 9 |
| | 9.11 Subgroup Analysis | 9 |
| | 9.12 Assessment of Site Homogeneity | 9 |
| Appen | ndix: Table Shells and List of Listings to be Generated | 9 |

This is the Statistical Analysis Plan (SAP) for the final analysis of data collected under Protocol NEU\_2017\_06. This SAP describes, in detail, the statistical methodology and statistical analyses for the above-mentioned protocol.

The original study protocol planned to continue study enrollment until 40 subjects were ablated (approximately 20 subjects ablated by interventional pulmonologists and 20 subjects ablated by thoracic surgeons) and completed Visit 3 (30 days  $\pm$  7 days after the first ablation procedure). However, study enrollment was temporarily halted after 10 subjects were enrolled to convene a meeting of the Data Safety Monitoring Board (DSMB) following the death of one subject. While the DSMB recommended that the study could continue enrollment, the decision was made to permanently stop study enrollment and follow the 10 previously-enrolled subjects through the end of the study follow-up period of 1 year post-ablation. As such, this decision impacts several of the analyses originally planned in the study protocol and those changes will be identified in the appropriate sections throughout this SAP.

### 1 Study Overview

#### 1.1 Study Objectives

The primary objective of the study was to evaluate the NeuWave Flex Microwave Ablation System in transbronchial ablation procedures for adult subjects with a medically inoperable primary soft tissue lesion, based on the following assessments:

- a. Device user experience survey
- b. Technical success
- c. Technique efficacy

Device user experience was collected from the treating physician who completed the User Experience Survey following each ablation procedure throughout the study, when applicable. The survey focused on procedure workflow and the user's assessment on ease/difficulty of using the device. The device user experience was designed to augment the Product Development Specialist's understanding of the usability of the Flex system and determine which enhancements, if any, are needed.

The secondary objectives were the following:

- 1. To evaluate safety through the monitoring of device-related and procedure-related adverse events (AEs) and all serious adverse events (SAEs), from start of ablation through 1-year post-ablation.
- 2. To establish device and procedure effectiveness by following subjects for 1-year postablation to ensure completeness and durability of treatment effect, based on standard endpoints in microwave ablation, as follows:
  - a. Primary efficacy rate
  - b. Secondary efficacy rate
  - c. Local soft lesion recurrence

- d. Length of hospital stay, measured from post-ablation to discharge
- e. Hospital readmission rate.
- 3. To calculate hospital readmission rate, defined as any readmission to the hospital within 30 days of the first ablation procedure (Visit 2A).

The exploratory objectives were the following:

- 1. To assess the quality of life post microwave ablation of the lung throughout the 1 year  $\pm$  1 month follow-up period.
- 2. To assess the level of pain during the initial 30 days  $\pm$  7 days post-ablation.

#### 1.2 Study Design

This was a prospective, multi-center, single-arm study for NEUWAVE Flex Microwave Ablation System in the ablation of soft tissue lesions of the lung for medically inoperable subjects, or those who elect not to have surgery. Prospective subjects were informed about the nature of the research, given the informed consent form (ICF) to read, and given the opportunity to ask any questions about the study. Once the subject understood the content of the ICF, s/he was asked to provide written consent. Individuals scheduled for microwave ablation of the lung were to be enrolled after providing informed consent and meeting study entry criteria, known as the inclusion and exclusion criteria. Subjects were to be followed for approximately 1 year following the first ablation procedure for safety and effectiveness outcomes.

## 2 Treatment Assignment

This was a single-arm study where all enrolled subjects underwent transbronchial microwave ablation with the NeuWave Flex Microwave Ablation System.

## 3 Randomization and Blinding Procedures

This was a single-arm, open-label study. No randomization occurred and no blinding procedures were required.

#### 4 Interval Windows

Interval windows are not defined for the purpose of analysis in this study outside of the visit windows that are provided in the Schedule of Assessments in Table 1 of the final protocol. There will be no assigning of observations to time points outside of the visit to which they are recorded in the electronic Case Report Forms (eCRFs). Data collected in Unscheduled Visit forms will be listed as such.

## 5 Levels of Significance

No hypotheses are specified for this study and no p-values are being calculated. Therefore, no level of significance is specified. All estimation of endpoints will be performed using 95% confidence intervals.

## 6 Analysis Sets

The study protocol identified two analysis sets:

- The Full Analysis Set (FAS) will consist of all subjects who are enrolled in the study and receive ablation through the flexible probe. The FAS was planned to be the primary analysis set for safety and effectiveness endpoints.
- The Per Protocol (PP) Analysis Set will consist of all subjects who are enrolled in the study
  and receive ablation through the flexible probe and have no major protocol deviations.
  Effectiveness analyses were planned to be repeated for the Per Protocol Set.

Given the decision to stop study enrollment at 10 subjects, only the Full Analysis Set will be defined for summarizing effectiveness and safety data in this study. A Per Protocol Analysis Set will not be defined.

## 7 Sample Size Justification

No formal hypotheses were planned to be tested in this study, and hence, a target sample size of 40 subjects (with an approximate equal distribution of device use by interventional pulmonologists and thoracic surgeons) was deemed adequate for a preliminary investigation of the feasibility of this procedure, as well as for providing sufficient information for appropriately sizing a subsequent study.

From a safety perspective, the AEs of interest in this study included: pneumothorax (requiring tube drainage), hemorrhage (bleeding requiring medical intervention), post-ablation syndrome, pain, pleural effusion (requiring tube drainage), infection, pneumonia, abscess, and bronchopleural fistula. A target sample size of 40 subjects provided a high likelihood of observing events in this composite and would allow for an initial evaluation of the frequency of occurrence relative to published literature in similar procedures.

As stated earlier, enrollment was stopped after 10 subjects received ablation and the original planned target of 40 subjects was not achieved.

## 8 Data Safety Monitoring Board

A DSMB was appointed by the Sponsor to review, on a regular basis, safety data from the study. The DSMB was to advise the Sponsor regarding the continuing safety of subjects and those yet to

be recruited to the study. Based on accumulating data from the study, the DSMB was to recommend whether to continue, suspend, modify, or stop the study. The composition, responsibilities, frequency of DSMB meetings, handling of emergency situations, and documentation of DSMB meetings was specified in the DSMB Charter and proceedings from DSMB meetings are maintained with the Sponsor.

### 9 Analyses to be Conducted

#### 9.1 General Conventions

Subject data will be summarized using listings and tables. All eCRF data will be listed per subject for all subjects. Descriptive statistical analyses will be provided for pre-specified study endpoints. Summaries for continuous variables will include number of observations (n), mean, standard deviation, median, minimum, and maximum. Summaries for categorical variables will include number and percentage.

Analyses will be conducted using SAS software version 9.4 or higher. During the course of analysis programming of tables that are mocked up in this SAP, minor modifications may become necessary. Examples of these minor modifications include, but are not limited to, re-wording of a footnote, addition of a footnote, re-labeling of a column, or addition or removal of a column from a listing. In cases where modifications to tables or listings are not related to a change in statistical analysis methodology or conclusions that could be made on the originally proposed methodology, then no amendment of the SAP is necessary. Any final analyses that differ from what has been specified in this document will be identified within the final statistical output and documented within the clinical study report.

#### 9.2 Disposition of Study Subjects

Subject disposition will be summarized in total using counts and percentages. The number and percentage of subjects completed and discontinued will be tabulated along with the specific reasons for discontinuation.

#### 9.3 Demographic, Baseline, and Subject Health Status Characteristics

Summary statistics of subject demographics and baseline characteristics (age, gender, childbearing potential, race, ethnicity, and body mass index) will be presented in total for the Full Analysis Set. Subject medical history will be summarized by Medical Dictionary for Regulatory Activities (MedDRA) system organ class and preferred term.

#### 9.4 Primary Endpoint Analyses

Device user experience feedback was collected from the treating physician who were to complete the User Experience Survey following each ablation procedure. The questionnaire was focused on procedure workflow and the user's assessment on ease/difficulty of using the device. Per the study

protocol, summary statistics were to be provided for each question in the survey; however, given the overall reduced sample size, only responses to the Probe Placement, Ablation Procedure, and General System Feedback sections will be summarized. All data collected on the User Experience Survey will be listed.

The number and percentage of subjects achieving technical success will be summarized and an exact 95% confidence interval will be presented. A similar summary will be presented for technique efficacy.

#### 9.5 Secondary Endpoint Analyses

The study protocol indicates that summaries will be provided for the primary and secondary efficacy rates as well as hospital readmission rates. However, data relevant to these endpoints will only be listed given the reduction in overall sample size. The number and percentage of subjects experiencing target lesion recurrence at any time during following will be summarized and an exact 95% confidence interval will be estimated, but the Kaplan-Meier analysis described in the study protocol will not be performed.

#### 9.6 Safety Analyses

Safety will be assessed through the incidence of AEs and SAEs, which will be coded using MedDRA. The number and percentage of subjects reporting AEs and SAEs will be summarized at the MedDRA system organ class and preferred term level. Similar summaries will also be provided for AEs and SAEs related to the study device, as well as for AEs and SAEs related to the study procedure. Related events are those where the relationship is indicated as Unlikely, Possibly, Probably, or Causal. Summaries of all AEs and SAEs reported within the first 30 days after the initial ablation procedure will be generated. All reported adverse events will be listed.

#### 9.7 Additional Endpoint Analyses

Counts and percentages will be provided for subject performance status as measured by the Eastern Cooperative Oncology Group (ECOG) classification at each visit. Summary statistics will be provided for the numeric pain rating scale measurement and hematology parameters at each visit. Pulmonary function tests will be summarized with summary statistics at each visit where they are measured and the change from the Screening visit measurement will also be summarized. Responses to each question of the EORTC QLQ-LC 13 will be summarized at each visit where the questionnaire was administered. Responses to the EORTC QLQ-C 30 will be listed.

Target lesion details including lesion type, lesion sub-type, size (largest and smallest diameter), location, distance from pleura, and shape will be summarized with statistics appropriate for categorical or continuous variables. Non-target lesion data will be listed. Selected information from the ablation procedure (duration of procedure, duration of ablation delivery, type of anesthesia, maximum power applied, and maximum temperature observed) will also be summarized with statistics appropriate for categorical or continuous variables.

Summary statistics will be presented for evaluations made by the independent reviewer for selected fields relating to ablation of the target lesion (largest diameter, smallest diameter, lesion location, distance from pleura, ablation margin, technical success, technique efficacy, and target lesion recurrence at any visit). All other target lesion data and all non-target lesion data from the independent reviewer will be listed.

#### 9.8 Plans for Interim Analysis

No formal interim analyses were planned or performed for this study outside of the data reviews that were pre-specified per the DSMB charter.

#### 9.9 Handling of Missing Data

All summaries will be performed only on subjects who receive ablation through the flexible probe. There will be no imputation of data for early terminated subjects or for missing data within the database.

#### 9.10 Sensitivity Analyses

No sensitivity analyses were planned per the study protocol given the absence of any hypotheses to be tested in this descriptive study and none will be performed.

#### 9.11 Subgroup Analysis

No subgroup analyses are planned for this study.

#### 9.12 Assessment of Site Homogeneity

No summaries or adjustments by study site are planned for this study.

## Appendix: Table Shells and List of Listings to be Generated

Table shells are provided, below, for all summaries to be generated for this study. Additionally, a list of all listings to be created is provided corresponding to the eCRFs that were used during this study. All fields collected will be listed.

NeuWave Medical, Inc. Protocol Number: NEU\_2017\_06

Page x of y

Program Name: XXXXXXXX.sas Run Date: mm/dd/yyyy hh:mm Data Last Modified: mm/dd/yyyy hh:mm

Table 1 Subject Disposition All Subjects

| | Total |
|-----------------------------|------------|
| Signed Informed Consent | XX |
| Full Analysis Set | xx (xx.x%) |
| Completed the Study | xx (xx.x%) |
| Discontinued from the Study | xx (xx.x%) |
| Reason for Discontinuation | |
| Withdrawal of consent | xx (xx.x%) |
| Surgical | xx (xx.x%) |
| Adverse Event | xx (xx.x%) |
| Death | xx (xx.x%) |
| Lost to Follow-up | xx (xx.x%) |
| Physician Decision | xx (xx.x%) |
| Other | xx (xx.x%) |

Note: All percentages are based on the number of subjects in the Full Analysis Set as the denominator.

Programming note: Only discontinuation reasons actually observed are to be displayed. Full Analysis Set includes all subjects who have a non-missing date of ablation on the Ablation Procedure CRF. >>

NeuWave Medical, Inc. Protocol: NEU\_2017\_06 

Program Name: XXXXXXXX.sas Run Date: mm/dd/yyyy hh:mm Data Last Modified: mm/dd/yyyy hh:mm

Table 2 Subject Demographics and Vital Signs Full Analysis Set

| Characteristics | Overall (N = ##) |
|-------------------------------------------|------------------|
| Race | |
| White | xx (xx.x%) |
| Black or African American | xx (xx.x%) |
| American Indian or Alaska Native | xx (xx.x%) |
| Native Hawaiian or Other Pacific Islander | xx (xx.x%) |
| Asian | xx (xx.x%) |
| Other | xx (xx.x%) |
| Ethnicity | |
| Hispanic or Latino | xx (xx.x%) |
| Not Hispanic or Latino | xx (xx.x%) |
| Not reported | xx (xx.x%) |
| Age (years) | |
| n | XX |
| Mean | XX.X |
| Standard Deviation | X.XXX |
| Median | XX.X |
| Minimum, Maximum | XX.X, XX.X |
| Gender | |
| Male | xx (xx.x%) |
| Female | xx (xx.x%) |
| Childbearing Potential | |
| Of childbearing potential | xx (xx.x%) |
| Permanently sterilized | xx (xx.x%) |
| Postmenopausal | xx (xx.x%) |
| Body Mass Index (kg/m2) | |
| n | XX |
| Mean | XX.X |
| Standard Deviation | X.XXX |
| Median | XX.X |
| Minimum, Maximum | XX.X, XX.X |

Programming note: Percentages for childbearing potential are based on the number of females in the study.

Program Name: XXXXXXXX.sas Run Date: mm/dd/yyyy hh:mm Data Last Modified: mm/dd/yyyy hh:mm

Table 3 Protocol Deviations Full Analysis Set

| Characteristics | Overall (N = ##) |
|---|---|
| Total Number of Protocol Deviations | xxx |
| Specific Types of Protocol Deviations [1] | |
| Informed Consent Process | xx (xx.x%) |
| Inclusion/Exclusion Criteria | xx (xx.x%) |
| Study Procedure | xx (xx.x%) |
| Visit Out of Window | xx (xx.x%) |
| Other | xx (xx.x%) |
| Sponsor Assessment of Protocol Deviations [1] | |
| Minor | xx (xx.x%) |
| Major | xx (xx.x%) |
| Number (%) of Subjects With at Least 1 Protocol Deviation [2] | xx (xx.x%) |

Denominator used is the total number of protocol deviations reported.
 Denominator used is the total number of subjects in the column header.

Program Name: XXXXXXXX.sas Run Date: mm/dd/yyyy hh:mm Data Last Modified: mm/dd/yyyy hh:mm

Table 4 Medical History by System Organ Class and Preferred Term Full Analysis Set

| System Organ Class | Preferred Term | Overall<br>(N = ##) |
|---|---|---|
| Total | | xx (xx.x%) |
| System Organ Class 1 | Preferred Term 1<br>Preferred Term 2<br>Preferred Term 3 | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) |
| System Organ Class 2 | Preferred Term 1<br>Preferred Term 2 | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) |
| System Organ Class 3 | Preferred Term 1<br>Preferred Term 2<br>Preferred Term 3 | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) |
| System Organ Class 4 | Preferred Term 1<br>Preferred Term 2 | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) |

Run Date: mm/dd/yyyy hh:mm Data Last Modified: mm/dd/yyyy hh:mm

Program Name: XXXXXXXX.sas

Table 5 ECOG Performance Status Over Time Full Analysis Set

| ECOG Score | Visit 1/<br>Screening | Visit 2A/<br>Day 0 | Visit 3/<br>Day 30 | Visit 4/<br>Month 6 | Visit 5/<br>Month 12 |
|---|---|---|---|---|---|
| 0 – Fully active | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 1 – Restricted in physically strenuous activity 2 – Ambulatory, capable of self care, unable to work | xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%) |
| 3 – Capable of only limited self care | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 4 – Completely disabled | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Programming note: The number of observed responses at each time point are summarized. No imputation will be performed for subjects not responding at a given visit. >>>

Program Name: XXXXXXXX.sas Run Date: mm/dd/yyyy hh:mm Data Last Modified: mm/dd/yyyy hh:mm

#### Table 6 Target Lesion Details – Visit 2A/Day 0 Full Analysis Set

| Characteristics | Overall (N = ##) |
|--------------------------------------------|------------------|
| Lesion Type | |
| NSCLC medically inoperable | xx (xx.x%) |
| NSCLC medically operable; declined surgery | xx (xx.x%) |
| Other | xx (xx.x%) |
| Lesion Sub-type | |
| Squamous cell carcinoma | xx (xx.x%) |
| Adenocarcinoma | xx (xx.x%) |
| Large cell carcinoma | xx (xx.x%) |
| Other | xx (xx.x%) |
| Lesion Location | |
| RUL | xx (xx.x%) |
| RML | xx (xx.x%) |
| RLL | xx (xx.x%) |
| LUL | xx (xx.x%) |
| LLL | xx (xx.x%) |
| Other | xx (xx.x%) |
| Lesion Shape | |
| Sphere | xx (xx.x%) |
| Ellipse | xx (xx.x%) |
| Triangular | xx (xx.x%) |
| Multilobar | xx (xx.x%) |
| Other | xx (xx.x%) |
| Distance from Pleura (cm) | |
| n | XX |
| Mean | XX.X |
| Standard Deviation | X.XXX |
| Median | XX.X |
| Minimum, Maximum | xx.x, xx.x |
| Largest Diameter (cm) | |
| n | XX |
| Mean | XX.X |
| Standard Deviation | X.XXX |
| Median | XX.X |
| Minimum, Maximum | XX.X, XX.X |

Program Name: XXXXXXXX.sas Run Date: mm/dd/yyyy hh:mm
Data Last Modified: mm/dd/yyyy hh:mm

# Table 6 Target Lesion Details – Visit 2A/Day 0 Full Analysis Set

| Characteristics | Overall (N = ##) |
|-------------------------------|------------------|
| Smallest Diameter (cm) | |
| n | XX |
| Mean | XX.X |
| Standard Deviation | X.XXX |
| Median | XX.X |
| Minimum, Maximum | XX.X, XX.X |
| Technical Success | |
| Yes | xx (xx.x%) |
| 95% Exact Confidence Interval | xx.x%, xx.x% |


Program Name: XXXXXXXX.sas Run Date: mm/dd/yyyy hh:mm Data Last Modified: mm/dd/yyyy hh:mm

## Table 7 Ablation Procedure Details Full Analysis Set

| Characteristics | Overall (N = ##) |
|-----------------------------------------|------------------|
| | (-,, |
| Type of Anesthesia | |
| General | xx (xx.x%) |
| Conscious sedation | xx (xx.x%) |
| Deep conscious sedation | xx (xx.x%) |
| Maximum Power Applied (watts) | |
| n | XX |
| Mean | XX.X |
| Standard Deviation | x.xxx |
| Median | XX.X |
| Minimum, Maximum | XX.X, XX.X |
| Maximum Temperature Observed (Celsius) | |
| n | XX |
| Mean | XX.X |
| Standard Deviation | x.xxx |
| Median | XX.X |
| Minimum, Maximum | XX.X, XX.X |
| Duration of Procedure (minutes) | |
| n | XX |
| Mean | XX.X |
| Standard Deviation | x.xxx |
| Median | XX.X |
| Minimum, Maximum | XX.X, XX.X |
| Duration of Ablation Delivery (minutes) | |
| n | xx |
| Mean | XX.X |
| Standard Deviation | x.xxx |
| Median | XX.X |
| Minimum, Maximum | xx.x, xx.x |
| Device Used | |
| Flex 6 Probe | xx (xx.x%) |
| Flex 4 Probe | xx (xx.x%) |

Program Name: XXXXXXXX.sas Run Date: mm/dd/yyyy hh:mm Data Last Modified: mm/dd/yyyy hh:mm

Table 7
Ablation Procedure Details
Full Analysis Set

| | Overall |
|---------------------------------------------|------------|
| Characteristics | (N = ##) |
| Final Ablation Zone, smallest diameter (cm) | |
| n | XX |
| Mean | XX.X |
| Standard Deviation | X.XXX |
| Median | XX.X |
| Minimum, Maximum | XX.X, XX.X |
| Total Number of Probe Repositions | |
| n | XX |
| Mean | XX.X |
| Standard Deviation | X.XXX |
| Median | XX.X |
| Minimum, Maximum | XX.X, XX.X |

NeuWave Medical, Inc. Protocol: NEU\_2017\_06 SAP Version 1.0: 29JAN2020 

Program Name: XXXXXXXX.sas Run Date: mm/dd/yyyy hh:mm Data Last Modified: mm/dd/yyyy hh:mm

## Table 8 Technique Efficacy and Target Lesion Recurrence Full Analysis Set

| Characteristics | Overall (N = ##) |
|---|---|
| Technique Efficacy at Day 30<br>Yes<br>95% Exact Confidence Interval | xx (xx.x%)<br>xx.x%, xx.x% |
| Target Lesion Recurrence Day 30 Through Month 12<br>Yes<br>95% Exact Confidence Interval | xx (xx.x%)<br>xx.x%, xx.x% |


Program Name: XXXXXXXX.sas Run Date: mm/dd/yyyy hh:mm Data Last Modified: mm/dd/yyyy hh:mm

Table 9 User Experience Survey Full Analysis Set

| Characteristics | Overall (N = ##) |
|---|---|
| Able to Pass Flex Probe through EWC as Expected | |
| Yes | xx (xx.x%) |
| No | xx (xx.x%) |
| Time to Place Probe in Acceptable Position (minutes) | |
| n | XX |
| Mean | XX.X |
| Standard Deviation | X.XXX |
| Median | XX.X |
| Minimum, Maximum | xx.x, xx.x |
| Number of 3D Scans for Probe Placement | |
| n | XX |
| Mean | XX.X |
| Standard Deviation | X.XXX |
| Median | XX.X |
| Minimum, Maximum | XX.X, XX.X |
| Distance From Probe to Center of Lesion (mm) | |
| n | XX |
| Mean | XX.X |
| Standard Deviation | X.XXX |
| Median | XX.X |
| Minimum, Maximum | XX.X, XX.X |
| Probe Repositioned After Initial Ablation for More Ablation | |
| Yes | xx (xx.x%) |
| No | xx (xx.x%) |
| Performing Ablation With NeuWave Flex System is Predictable | |
| 1 – Disagree | xx (xx.x%) |
| 2 | xx (xx.x%) |
| 3 | xx (xx.x%) |
| 4 | xx (xx.x%) |
| 5 - Agree | xx (xx.x%) |

Program Name: XXXXXXXX.sas Run Date: mm/dd/yyyy hh:mm Data Last Modified: mm/dd/yyyy hh:mm

Table 9 User Experience Survey Full Analysis Set

| | Overall |
|---|---|
| Characteristics | (N = ##) |
| Ablation With NeuWave Flex System is Simple to Use | |
| 1 – Disagree | xx (xx.x%) |
| 2 | xx (xx.x%) |
| 3 | xx (xx.x%) |
| 4 | xx (xx.x%) |
| 5 - Agree | xx (xx.x%) |
| Technical Success can be Achieved Similar to a Percutaneous Approach | |
| 1 – Disagree | xx (xx.x%) |
| 2 | xx (xx.x%) |
| 3 | xx (xx.x%) |
| 4 | xx (xx.x%) |
| 5 - Agree | xx (xx.x%) |
| Confidently Locate the Probe and Targeted Lesion Using my Imaging Tool: | c |
| 1 – Disagree | xx (xx.x%) |
| 2 | xx (xx.x%) |
| 3 | xx (xx.x%) |
| 4 | xx (xx.x%) |
| 5 - Agree | xx (xx.x%) |
| | , , |
| Confidently Locate the Ablation Zone Created During Flex Ablation Proceed | |
| 1 – Disagree | xx (xx.x%) |
| 2 | xx (xx.x%) |
| 3 | xx (xx.x%) |
| 4 | xx (xx.x%) |
| 5 – Agree | xx (xx.x%) |

NeuWave Medical, Inc. Protocol: NEU\_2017\_06 SAP Version 1.0: 29JAN2020 

Program Name: XXXXXXXX.sas Run Date: mm/dd/yyyy hh:mm Data Last Modified: mm/dd/yyyy hh:mm


Table 10 Pulmonary Function Tests and Change From Screening Over Time Full Analysis Set

| Parameter | Visit 1/ | Visit 4/ | Change From | Visit 5/ | Change From |
|---|---|---|---|---|---|
| Statistic | Screening | Month 6 | Visit 1 to Visit 4 | Month 12 | Visit 1 to Visit |
| FeNO (ppb) | | | | | |
| n | xx | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| Standard Deviation | x.xxx | X.XXX | X.XXX | X.XXX | X,XXX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Minimum, Maximum | XX.X, XX.X | xx.x, xx.x | xx.x, xx.x | XX.X, XX.X | xx.x, xx.x |
| DLCO (mL/min/mmHg) | | | | | |
| n | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| Standard Deviation | X.XXX | X.XXX | X.XXX | X.XXX | X.XXX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Minimum, Maximum | XX.X, XX.X | xx.x, xx.x | xx.x, xx.x | XX.X, XX.X | xx.x, xx.x |
| DLCO (%) | | | | | |
| SpO2 (%) | | | | | |
| FVC (mL) | | | | | |
| EVO (0/) | | | | | |

FVC (%)

FEV1 (mL)

FEV1 (% of predicted)

FEV1/FVC (% of predicted)

Plethysmographic TLC (mL)

Plethysmographic TLC (% of predicted)

Plethysmographic FRC (mL)

Plethysmographic FRC (% of predicted)
Gas Dilution TLC (mL)

Gas Dilution TLC (% of predicted)

Gas Dilution FRC (mL)

Gas Dilution FRC (% of predicted)

<>> Programming note: The number of observed responses at each time point are summarized. No imputation will be performed for subjects not responding at a given visit. >>>

NeuWave Medical, Inc. Protocol: NEU\_2017\_06

Program Name: XXXXXXXX.sas Run Date: mm/dd/yyyy hh:mm Data Last Modified: mm/dd/yyyy hh:mm

Table 11 Hematology Tests Over Time Full Analysis Set

| Parameter | Visit 1/ | Visit 3/ | Visit 4/ | Visit 5/ |
|---|---|---|---|---|
| Statistic | Screening | Day 30 | Month 6 | Month 12 |
| RBC (M/uL) | | | | |
| n | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X |
| Standard Deviation | X.XXX | X.XXX | X.XXX | X.XXX |
| Median | XX.X | XX.X | XX.X | XX.X |
| Minimum, Maximum | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| WBC (K/uL) | | | | |
| n | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X |
| Standard Deviation | X.XXX | X.XXX | X.XXX | X.XXX |
| Median | XX.X | XX.X | XX.X | XX.X |
| Minimum, Maximum | XX.X, XX.X | XX.X, XX.X | xx.x, xx.x | XX.X, XX.X |
| Neutrophils (%) | | | | |
| Lymphocytes (%) | | | | |
| Monocytes (%) | | | | |
| Eosinophils (%) | | | | |
| Basophils (%) | | | | |
| Hemoglobin (g/dL) | | | | |
| Hematocrit (%) | | | | |
| Mean Corpuscular Volume (fL) | | | | |
| Platelet Count (K/uL) | | | | |
| PTA (%) | | | | |
| APTT (seconds) | | | | |
| PT (seconds) | | | | |
| INR (ratio) | | | | |

NeuWave Medical, Inc. Protocol: NEU\_2017\_06 SAP Version 1.0: 29JAN2020 

<sup>&</sup>lt;<< Programming note: The number of observed responses at each time point are summarized. No imputation will be performed for subjects not responding at a given visit. >>>

Program Name: XXXXXXXX.sas Run Date: mm/dd/yyyy hh:mm Data Last Modified: mm/dd/yyyy hh:mm

Table 12 Numeric Pain Rating Scale Over Time Full Analysis Set

| Parameter | Visit 1/ | Visit 2A/ | Visit 2B/ | Visit 3/ |
|---|---|---|---|---|
| Statistic | Screening | Day 0 | Day 1 | Day 30 |
| Self-Reported Pain Intensity in the Last 24 Hours | | | | |
| n | XX | Xx | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X |
| Standard Deviation | X.XXX | X.XXX | X.XXX | X.XXX |
| Median | XX.X | XX.X | XX.X | XX.X |
| Minimum, Maximum | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |

Note: A pain score of 0 indicates no pain, 5 indicates moderate pain, and 10 indicates worst possible pain.

Program Name: XXXXXXXX.sas Run Date: mm/dd/yyyy hh:mm Data Last Modified: mm/dd/yyyy hh:mm

Table 13 EORTC QLQ-LC 13 Full Analysis Set

| Characteristics | Visit 1/<br>Screening<br>(N = ##) | Visit 2A/<br>Day 0<br>(N = ##) | Visit 2B/<br>Day 1<br>(N = ##) | Visit 3/<br>Day 30<br>(N = ##) | Visit 4/<br>Month 6<br>(N = ##) | Visit 5/<br>Month 12<br>(N = ##) |
|---|---|---|---|---|---|---|
| How much did you cough? | | | | | | |
| Not at all | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| A little | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Quite a bit | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Very much | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| No response | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Did you cough up blood? | | | | | | |
| Not at all | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| A little | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Quite a bit | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Very much | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| No response | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Were you short of breath when you rested?

Were you short of breath when you walked?

Were you short of breath when you climbed stairs?

Have you had a sore mouth or tongue?

Have you had trouble swallowing?

Have you had tingling hands or feet?

Have you had hair loss?

Have you had pain in your chest?

Have you had pain in your arm or shoulder?

Have you had pain in other parts of your body?

Did you take any medication for pain?

If yes, how much did it help?

Note: Responses given refer to during the past week.

Program Name: XXXXXXXX.sas Run Date: mm/dd/yyyy hh:mm Data Last Modified: mm/dd/yyyy hh:mm

Table 14 Adverse Events by System Organ Class and Preferred Term Full Analysis Set

| System Organ Class | Preferred Term | Overall<br>(N = ##) |
|---|---|---|
| Total | | xx (xx.x%) |
| System Organ Class 1 | Preferred Term 1<br>Preferred Term 2<br>Preferred Term 3 | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) |
| System Organ Class 2 | Preferred Term 1<br>Preferred Term 2 | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) |
| System Organ Class 3 | Preferred Term 1<br>Preferred Term 2<br>Preferred Term 3 | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) |
| System Organ Class 4 | Preferred Term 1<br>Preferred Term 2 | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) |


Program Name: XXXXXXXX.sas Run Date: mm/dd/yyyy hh:mm Data Last Modified: mm/dd/yyyy hh:mm

The following tables will have the same format as Table 14:

| Table 15 | Serious Adverse Events by System Organ Class and Preferred Term Full Analysis Set |
|---|---|
| Table 16 | Adverse Events Related to the Study Device by System Organ Class and Preferred Term Full Analysis Set |
| Table 17 | Serious Adverse Events Related to the Study Device by System Organ Class and Preferred Term Full Analysis Set |
| Table 18 | Adverse Events Related to the Study Procedure by System Organ Class and Preferred Term Full Analysis Set |
| Table 19 | Serious Adverse Events Related to the Study Procedure by System Organ Class and Preferred Term Full Analysis Set |
| Table 20 | Adverse Events Related to the Study Device Within 30 Days of the Initial Ablation Procedure by System Organ Class and Preferred Term Full Analysis Set |
| Table 21 | Serious Adverse Events Related to the Study Device Within 30 Days of the Initial Ablation Procedure by System Organ Class and Preferred Term Full Analysis Set |

Program Name: XXXXXXXX.sas Run Date: mm/dd/yyyy hh:mm Data Last Modified: mm/dd/yyyy hh:mm

Table 22 Target Lesion Details – Independent Reviewer Full Analysis Set

| | Overall |
|-----------------------------------------|------------|
| Characteristics | (N = ##) |
| Lesion Location | |
| RUL | xx (xx.x%) |
| RML | xx (xx.x%) |
| RLL | xx (xx.x%) |
| LUL | xx (xx.x%) |
| LLL | xx (xx.x%) |
| Other | xx (xx.x%) |
| Distance from Pleura (cm) | |
| n | XX |
| Mean | XX.X |
| Standard Deviation | x.xxx |
| Median | XX.X |
| Minimum, Maximum | XX.X, XX.X |
| T (D) | |
| Largest Diameter (cm) | |
| n | XX |
| Mean | XX.X |
| Standard Deviation | X.XXX |
| Median | XX.X |
| Minimum, Maximum | XX.X, XX.X |
| Smallest Diameter (cm) | |
| n | xx |
| Mean | XX.X |
| Standard Deviation | X.XXX |
| Median | XX.X |
| Minimum, Maximum | XX.X, XX.X |
| Ablation Margin, Smallest Diameter (cm) | |
| n<br>M | XX |
| Mean | XX.X |
| Standard Deviation | X.XXX |
| Median | XX.X |
| Minimum, Maximum | XX.X, XX.X |

Program Name: XXXXXXXX.sas Run Date: mm/dd/yyyy hh:mm Data Last Modified: mm/dd/yyyy hh:mm

Table 22 Target Lesion Details – Independent Reviewer Full Analysis Set

| Characteristics | Overall (N = ##) |
|---------------------------------------------|------------------|
| Technical Success – Visit 2A/Day 0 | |
| Yes | xx (xx.x%) |
| 95% Exact Confidence Interval | xx.x%, xx.x% |
| Technique Efficacy at Day 30 | |
| Yes | xx (xx.x%) |
| 95% Exact Confidence Interval | xx.x%, xx.x% |
| Target Lesion Recurrence Day 30 to Month 12 | |
| Yes | vv (vv v0/) |
| 100 | xx (xx.x%) |
| 95% Exact Confidence Interval | xx.x%, xx.x% |


Program Name: XXXXXXXX.sas Run Date: mm/dd/yyyy hh:mm Data Last Modified: mm/dd/yyyy hh:mm

The following listings will be generated for this study:

| Listing 1 | Inclusion/Exclusion Criteria |
|------------|-----------------------------------------------|
| | All Subjects |
| Listing 2 | Inclusion/Exclusion Criteria – Ablation Visit |
| | All Subjects |
| Listing 3 | Study Visits |
| | All Subjects |
| Listing 4 | Study Visit Details |
| | All Subjects |
| Listing 5 | Demographics |
| | All Subjects |
| Listing 6 | Pregnancy Test |
| | All Subjects |
| Listing 7 | Medical History |
| | All Subjects |
| Listing 8 | Surgical History |
| | All Subjects |
| Listing 9 | Radiation History |
| | All Subjects |
| Listing 10 | Vital Signs |
| | All Subjects |
| Listing 11 | ECOG Performance Status |
| | All Subjects |
| Listing 12 | Pain Rating Scale (NPRS) |
| | All Subjects |
| Listing 13 | Pulmonary Function Tests |
| | All Subjects |
| Listing 14 | Hematology |
| | All Subjects |
| Listing 15 | Genetic Markers Testing |
| | All Subjects |

NeuWave Medical, Inc. Protocol: NEU\_2017\_06 SAP Version 1.0: 29JAN2020 

Program Name: XXXXXXXX.sas Run Date: mm/dd/yyyy hh:mm Data Last Modified: mm/dd/yyyy hh:mm

| Listing 16 | EORTC QLQ-C 30 |
|------------|--------------------------------------------|
| | All Subjects |
| Listing 17 | EORTC QLQ-LC 13 |
| | All Subjects |
| Listing 18 | Target Lesion Details |
| | All Subjects |
| Listing 19 | Non-Target Lesion Details |
| | All Subjects |
| Listing 20 | Target Lesion Details Central Reviewer |
| | All Subjects |
| Listing 21 | Non-Target Lesion Details Central Reviewer |
| | All Subjects |
| Listing 22 | Ablation Procedure |
| | All Subjects |
| Listing 23 | Imaging |
| | All Subjects |
| Listing 24 | User Experience Survey |
| | All Subjects |
| Listing 25 | Discharge |
| | All Subjects |
| Listing 26 | UB-04 |
| | All Subjects |
| Listing 27 | Concomitant Procedures |
| | All Subjects |
| Listing 28 | Concomitant Medications |
| | All Subjects |
| Listing 29 | Adverse Events |
| | All Subjects |
| Listing 30 | Protocol Deviations |
| | All Subjects |
| Listing 31 | Death |
| | All Subjects |

Program Name: XXXXXXXX.sas Run Date: mm/dd/yyyy hh:mm Data Last Modified: mm/dd/yyyy hh:mm

| Listing 32 | Subject Completion/Discontinuation |
|------------|------------------------------------|
| | All Subjects |